CLINICAL TRIAL: NCT05129059
Title: The Effect of Logotherapy Counseling Programme on Dignity and Chronic Sorrow in Palliative Care Patients Experiencing Chronic Sorrow
Brief Title: Logotherapy Counseling Programme for Palliative Care Patients With Chronic Sorrow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yasemin Eskigülek, RN, MSN, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA21/276
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Palliative Care; Cancer
Keywords: logotherapy; nursing; meaning in life; chronic sorrow; dignity
MeSH Terms: conditions — Neoplasms | interventions — Logotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Logotherapy (Experimental): Participants will receive individual logotherapy counseling by the investigator for 8 visits in 4 weeks.
  Interventions: Other: Logotherapy
- Control (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Other: Logotherapy — Logotherapy is a method of finding meaning with three basic principles. The first principle is that life is meaningful in every situation , even in the most desperate moments. The second principle is that the main source of motivation is the desire to find meaning in life. The third is that an individual is free to choose his own attitude even in the worst conditions.
  Arms: Logotherapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of logotherapy counseling program on chronic sorrow, meaning of life and dignity of palliative care patients.

DETAILED DESCRIPTION:
Palliative care patients experience psychosocial and spiritual problems such as depressed mood, fear of metastasis, uncertainty, lack of pleasure, fear of suffering, and chronic sorrow. Logotherapy is a meaning-centered intervention helping the individual to discover the meaning of life and increasing the spiritual well-being and quality of life of the individual. In this study, the effect of logotherapy counseling program on dignity, chronic sorrow and meaning of life of palliative care patients will be evaluated.

In this study, the participants will be randomized in a single blind manner (participant) to either intervention (8 session-4 week logotherapy) or control (routine care) groups.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients due to advanced cancer Patients informed of cancer diagnosis at least 1 month Patients reporting to have chronic sorrow Patients with palliative performance scale score at least 50% Patients having life expectancy more than 6 months Patients who volunteered to participate in the study and signed written informed consent

Exclusion Criteria:

Clinically diagnosed mental disorder Patients with palliative performance scale score < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
meaning in life | baseline and 8 weeks
  Meaning in life scale is a validated, 7-points Likert type scale with 2 dimensions. Possible scores range from 5 to 35 for each dimensions. Change= score of present meaning subscale> searched meaning subscale (8 week subscale-baseline subscale
dignity | baseline and 8 weeks
  The Patient Dignity Inventory is a valid, 5-points Likert type scale with 5 dimensions. Possible scores range from 25-125. Change= Lower score from the patient dignity inventory at the end of intervention compared to baseline.
chronic sorrow | baseline and 8 weeks
  Prolonged grief disorder scale-patient form is a valid, 5-points Likert type scale. Possible scores range from 12 to 60. Change= Lower score from the scale at the end of intervention compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Eskigülek, Principal Investigator — Baskent University; Sultan Kav, Study Director — Baskent University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eskigulek Y, Kav S. Effect of logotherapy counseling program on chronic sorrow, dignity, and meaning in life of palliative care patients: a randomized controlled trial. Support Care Cancer. 2024 Aug 13;32(9):587. doi: 10.1007/s00520-024-08792-w. PMID 39138762